CLINICAL TRIAL: NCT00555178
Title: Regulatory T Cells (Tregs) in Polymorphic Light Eruption
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Peter Wolf, MD, Professor of Bioimmunotherapy, Medical University of Graz
Other Study IDs: 18-116 ex 06/07
Record Dates: First submitted 2007-11-07; First posted 2007-11-08 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: Polymorphic Light Eruption; Psoriasis; Atopic Eczema
Keywords: Polymorphic light eruption; Regulatory T cells (Tregs); Seasonal fluctuation; UV radiation; Phototherapy
MeSH Terms: conditions — Psoriasis; Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: Patients with polymorphic light eruption without medical photohardening treatment
- 2: Patients with polymorphic light eruption treated with medical photohardening
- 3: Patients with other disorders (including psoriasis) treated with phototherapy
- 4: Normal healthy subjects

SUMMARY:
Polymorphic light eruption (PLE) is a photodermatosis with an extremely high prevalence, particularly among young women (up to 20%). The disease is characterized through itchy skin lesions on sun-exposed body sites occurring after sun exposure mostly in spring and early summer. Its etiopathogenesis is unknown but resistance to UV-induced immunosuppression with subsequent immune reactions against skin photoneoantigens has been suggested. Regulatory T cells (CD4+CD25+FoxP3+) (Tregs), a subset of T helper cells, are crucial for the induction of immunosuppression. We will test the hypothesis that PLE patients show pathogenic fluctuating Treg levels and function and related parameters over the seasons of the year, possibly being responsible for lack of immune modulation and autoimmunity in PLE. Natural or medical photohardening may normalize Treg deficiency in PLE and lead to clinical adaption in summer. Better insight into the pathogenesis of PLE may give clues to develop new therapeutic strategies.

DETAILED DESCRIPTION:
PLE patients will be recruited through the Photodermatology Unit of the Department of Dermatology, Medical University of Graz, Graz, Austria. Eligible patients will be identified through diagnosis-related computer-assisted search in the electronic patient chart system of the Unit. The diagnosis of PLE will be verified by patient's history, clinical symptoms, histologic findings, laboratory studies and/or phototesting procedures.

The levels and function of Tregs, memory T cells, neutrophils, mast cells, Langerhans cells, cytokine and chemokine profiles, vitamin D levels in the blood and/or skin will be studied in PLE patients compared to control groups. Volunteers of four groups will be enrolled in this study: i) patients with PLE undergoing preventive medical UV photohardening in spring; ii) PLE patients not undergoing preventive UV photohardening; iii) healthy control subjects; and iv) patients with other diseases (including psoriasis, atopic dermatitis, and other conditions) undergoing therapeutic phototherapy.

Blood will be taken by venous puncture (mainly of a cubital vein) from the individual study participants at four defined time points during the year: (i) spring (March to April) (before medical photohardening in PLE patients); (ii) spring/early summer (April to June) (immediately after medical photohardening of PLE patients); (iii) late summer (August to September); and (iv) late fall (November to December). In addition, optional skin biopsies will be taken to study the parameters listed above. The statistical power analysis (alpha 0.05; power 0.8; assumed difference in Treg level/function of 30% among groups; based on the data by Myara et al., 2005) revealed that 23 patients (21+2 expected drop-outs) need to be enrolled per patient group. All patients of the non-PLE groups will be sex- and age (plus/minus 5 years)-matched to the PLE subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years
* Patients with confirmed PLE diagnosis either by typical anamnesis and/or typical histology of lesions and/or positive phototesting results (group 1 and 2); healthy subjects (group 3); patients with phototherapy-responsive disease (including psoriasis, atopic dermatitis, and other conditions (group 4).
* Good general health status

Exclusion Criteria:

* Presence or history of malignant skin tumors
* Dysplastic melanocytic nevus syndrome
* Certain photosensitive disorders (including porphyria, chronic actinic dermatitis, Xeroderma pigmentosum, basal cell nevus syndrome)
* Autoimmune disease (lupus erythematodes, scleroderma, dermatomyositis)
* Systemic treatment with steroids and/or other immunosuppressive drugs within the last 6 months
* Antinuclear antibodies (ds-DNA, Ro, La)
* First-degree relatives of PLE patients (exclusion criterion for group 3 and 4
* Pregnancy and breastfeeding
* Ongoing or planned specific hyposensitization treatment (i.e. specific immunotherapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care clinic patients and community sample
Sampling Method: Non-Probability Sample
Enrollment: 92 (Estimated)
Dates: Start 2008-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Treg level and function | Prospective

SECONDARY OUTCOMES:
Blood and/or skin cytokine and chemokine levels, vitamin D status, and other immunoregulatory parameters (see above) | prospective

CONTACTS AND LOCATIONS:
Overall Officials: Peter Wolf, MD, Principal Investigator — Medical University of Graz
Locations (2):
- Austria (2):
  - Medical University of Graz, Department of Dermatology, Graz
  - Medical University of Graz, Graz